CLINICAL TRIAL: NCT00136825
Title: N-acetylcysteine as Treatment in Cocaine Addiction
Brief Title: Effectiveness of N-acetylcysteine in Treating Cocaine Dependent Individuals - 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-18501-1; F32-18501-1; DPMC
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2007-08

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine; treatment
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): Identical appearing placebo pill containing lactose powder, packaged to have similar odor as N-Acetylcysteine in capsule form
  Interventions: Drug: Placebo
- 1 (Experimental): N-Acetylcysteine
  Interventions: Drug: N-Acetylcysteine

INTERVENTIONS:
Drug: N-Acetylcysteine
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
Recent findings have suggested that N-acetylcysteine (NAC) substantially reduces cocaine drug-seeking behavior in formerly cocaine dependent rats. The purpose of this study is to determine the safety, tolerability, and cue reactivity effects of NAC in cocaine dependent individuals and non-dependent healthy controls.

DETAILED DESCRIPTION:
Recent findings have suggested that N-acetylcysteine (NAC) substantially reduces cocaine-primed drug-seeking behavior in formerly cocaine dependent rats. The purpose of this study is to determine the safety, tolerability, and cue reactivity effects of NAC in cocaine dependent individuals and non-dependent healthy controls.

Participants in this study will include 20 non-treatment seeking cocaine dependent individuals and 12 healthy, non-dependent controls. Participants will be recruited via word-of-mouth and advertisements. Cocaine dependent participants will undergo two 3-day hospital stays. Healthy controls will be followed throughout the study on an outpatient basis. All participants will be randomly assigned to receive either 600 mg of NAC or placebo. Medication or placebo will be administered twice each day. Participants will be evaluated for side effects throughout the study. After administration of the final dose of medication or placebo, participants will undergo cue reactivity testing. This will include a standardized protocol of slides demonstrating cocaine acquisition, use of cocaine, and cocaine-related paraphernalia. Before, during, and after cue reactivity procedures, standardized behavioral and cognitive scales will be used to assess cocaine craving, cocaine seeking, and subjective effects of the cocaine "high." The following week participants will be crossed over so that they will receive the other treatment. All study procedures will be performed a second time. Participants will be contacted during Week 3 in order to determine if any residual side effects or adverse events occurred from the medication and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Not seeking treatment for drugs of abuse
* Diagnostic and Statistical Manual of Mental Disorders-IV diagnosis of cocaine dependence (not applicable for individuals enrolling as healthy controls)
* Positive urine drug screen test for cocaine (not applicable for individuals enrolling as healthy controls)
* Females must use adequate forms of contraception throughout the study
* Stable residence for the 30 days prior to enrollment
* No history of N-acetylcysteine within the 7 days prior to enrollment
* Nicotine smokers staying at the inpatient unit must use the nicotine patch during inpatient stay

Exclusion Criteria:

* Dependence on any psychoactive substance other than alcohol, nicotine, or marijuana; control subjects cannot be dependent on cocaine
* Need for medication detoxification for alcohol
* History of psychiatric disorders, including depression, bipolar disorder, post traumatic stress disorder, dementia, and organic brain disorder
* Suicidal or homicidal behavior within the 30 days prior to enrollment
* History of psychotic symptoms, including those observed during cocaine use
* History of serious medical illness, including cardiovascular disease, angina, myocardial infarction, liver disease, and kidney disease
* History of neurologic, metabolic, neoplastic, nutritional, inflammatory, or endocrine disorders
* Court requirement to receive treatment
* Expecting elective surgery within the 5 weeks prior to enrollment
* Known hypersensitivity to N-acetylcysteine
* Use of antidepressants (such as selective serotonin reuptake inhibitors or tricyclics), dopamine agonists, or psychotropic medications (such as anticonvulsants, antipsychotics, anxiolytics, or psychostimulants) within the 14 days prior to enrollment
* Pregnant or breastfeeding
* History of asthma
* History of seizures
* Participation in treatment for cocaine abuse within the 30 days prior to enrollment
* Lactose intolerance

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2003-03; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Tolerability of N-Acetylcysteine | Measured throughout both inpatient stays

SECONDARY OUTCOMES:
Reactivity to pictures of cocaine | Measured after 4th and final dose of med/placebo during each hospital stay
Cocaine withdrawal | Measured at admission, then discharge, for each hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Steven D LaRowe, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] LaRowe SD, Mardikian P, Malcolm R, Myrick H, Kalivas P, McFarland K, Saladin M, McRae A, Brady K. Safety and tolerability of N-acetylcysteine in cocaine-dependent individuals. Am J Addict. 2006 Jan-Feb;15(1):105-10. doi: 10.1080/10550490500419169. PMID 16449100
- [Result] LaRowe SD, Myrick H, Hedden S, Mardikian P, Saladin M, McRae A, Brady K, Kalivas PW, Malcolm R. Is cocaine desire reduced by N-acetylcysteine? Am J Psychiatry. 2007 Jul;164(7):1115-7. doi: 10.1176/ajp.2007.164.7.1115. PMID 17606664